CLINICAL TRIAL: NCT01746420
Title: A Phase II Randomized, Single Ascending Dose, Double-blinded, Placebo Controlled, Multi-center Study of the Effects of rhPDGF-BB Injection on Lateral Epicondylitis
Brief Title: Phase II Study of the Effects of rhPDGF-BB Injection on Lateral Epicondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMimetic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMTI-2010-02
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Lateral Epicondylitis
Keywords: elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Becaplermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo Control (Placebo Comparator): Dose A - sodium acetate buffer (0 mg rhPDGF-BB)
  Interventions: Drug: Placebo
- 0.45 mg rhPDGF-BB (Experimental): Dose B - sodium acetate buffer + 0.45 mg rhPDGF-BB
  Interventions: Drug: rhPDGF-BB Injection
- 0.75 mg rhPDGF-BB (Experimental): Dose C - sodium acetate buffer + 0.75 mg rhPDGF-BB
  Interventions: Drug: rhPDGF-BB Injection
- 1.5 mg rhPDGF-BB (Experimental): Dose D - sodium acetate buffer + 1.5 mg rhPDGF-BB
  Interventions: Drug: rhPDGF-BB Injection
- 3.0 mg rhPDGF-BB (Experimental): Dose E - sodium acetate buffer + 3.0 mg rhPDGF-BB
  Interventions: Drug: rhPDGF-BB Injection

INTERVENTIONS:
Drug: rhPDGF-BB Injection — Comparison of placebo control (0 mg rhPDGF-BB) and different dosages (0.45, 0.75, 1.5, and 3.0 mg) of rhPDGF-BB Injection administered through a one-time injection
  Arms: 0.45 mg rhPDGF-BB; 0.75 mg rhPDGF-BB; 1.5 mg rhPDGF-BB; 3.0 mg rhPDGF-BB
Drug: Placebo — sodium acetate buffer (0 mg rhPDGF-BB)
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to determine whether recombinant human platelet-derived growth factor (rhPDGF-BB) Injection is effective in the treatment of lateral epicondylitis (tennis elbow).

DETAILED DESCRIPTION:
Methodology: Randomized, single ascending dose, double-blinded, placebo controlled, multi-center study

Study Center(s): 6

Number of Subjects: 100

Diagnosis and Main Inclusion Criteria: Lateral epicondylitis; male and female subjects 21 -80 years of age

Study Drug, Dose, Regimen:

Dose A: sodium acetate buffer alone - placebo control Dose B: sodium acetate buffer + 0.45 mg rhPDGF-BB Dose C: sodium acetate buffer + 0.75 mg rhPDGF-BB Dose D: sodium acetate buffer + 1.5 mg rhPDGF-BB Dose E: sodium acetate buffer + 3.0 mg rhPDGF-BB

Duration and Route of Administration: Single administration dose by injection into the extensor carpi radialis brevis (ECRB)

Duration of Follow-up: 24 weeks (6 months) post-operative follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed the Institutional Review Board (IRB) approved Informed Consent Form specific to this study prior to enrollment
2. Subject has a clinical diagnosis of lateral epicondylitis
3. Subject's symptoms can be reproduced with resisted supination or wrist dorsiflexion
4. Subject's symptoms have persisted for at least 3 months despite conservative treatment that includes one or combinations of:

   1. Physical therapy
   2. Splinting
   3. Nonsteroidal antiinflammatory drug (NSAID)
   4. Corticosteroid injection
5. Subject is independent, ambulatory, and can comply with all post-injection evaluations and visits
6. Subject is 21-80 years of age and considered to be skeletally mature

Exclusion Criteria:

1. Subject has undergone previous corticosteroid injection therapy to the effected elbow in less than three months prior to enrollment
2. Subject has received previous Platelet Rich Plasma (PRP) injection to the affected elbow
3. Subject is deemed to require a corticosteroid injection into the affected elbow during the course of the study
4. Subject uses chronic medications known to affect the skeleton (e.g. glucocorticoid usage >10mg/day)
5. Subject has undergone surgical intervention to the affected elbow for the treatment of lateral epicondylitis
6. Subject has a positive medical history of any of the following:

   1. medial epicondylitis
   2. radial tunnel syndrome
   3. carpal tunnel syndrome
   4. septic or gouty arthritis
   5. cervical radiculopathy
   6. trauma to the affected elbow within the past 6 weeks
   7. neuromuscular or musculoskeletal deficiency, which limits the ability to perform functional measurement (e.g. grip strength test)
7. Subject currently has an acute infection at the injection site
8. Subject has tested positive or been treated for a malignancy in the past or is suspected of having a malignancy or are currently undergoing radio- or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed rhPDGF-BB Injection treatment site
9. Subject is physically or mentally compromised (e.g. currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.) to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant
10. Subject has an allergy to yeast-derived products
11. Subject has received an investigational therapy or approved therapy for investigational use within 30 days of injection procedure or during the follow-up phase of this study
12. Subject is a prisoner, or is known or suspected to be transient
13. Subject's condition represents a worker's compensation case
14. Subject is currently involved in a health-related litigation procedure
15. Subject has documented evidence of a history (e.g. liver testing) of drug/alcohol abuse within the 12 months prior to screening for study entry
16. Subject is pregnant, or able to become pregnant but not practicing a medically-accepted form of birth control, and/or intending to become pregnant during this study period

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12-12 (Actual); Primary Completion 2014-10-21 (Actual); Study Completion 2014-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Akelman, MD, Principal Investigator — Brown University
Locations (6):
- United States (6):
  - Arizona Research Center, Phoenix, Arizona
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Coastal Orthopedics & Sports Medicine, Bradenton, Florida
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - OrthoCarolina, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Control: Dose A - sodium acetate buffer (0 mg rhPDGF-BB)
  rhPDGF-BB Injection: Comparison of placebo control (0 mg rhPDGF-BB) and different dosages (0.45, 0.75, 1.5, and 3.0 mg) of rhPDGF-BB Injection administered through a one-time injection
Period: Overall Study
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Started | 20 | 20 | 20 | 20 | 20
Completed | 17 | 18 | 17 | 20 | 20
Not Completed | 3 | 2 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 100
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 44.2 (7.1) | 49 (6.9) | 46 (7) | 47.4 (12.4) | 49 (8.3) | 47.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 8 | 10 | 9 | 51
  Male | 8 | 8 | 12 | 10 | 11 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 3 | 5
  White | 18 | 19 | 20 | 17 | 15 | 89
  More than one race | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Elbow Pain Assessments (VAS), Treated Subjects
Description: Subjects were asked to report current pain level at the fusion site on a 100 mm Visual Analog Scale (with 0 being no pain and 100 being worst pain imaginable).
Time Frame: Baseline, 2, 4, 8, 12, and 24 weeks
Population: Analysis conducted on patients at Baseline, 2, 4, 8, 12, and 24 weeks time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
score on a scale
  Baseline | 76.6 (14.4) | 77.7 (9.2) | 75.9 (16.9) | 72 (19.9) | 72.2 (20.6)
  Week 2: number analyzed (Participants) | 20 | 20 | 20 | 19 | 20
  Week 2 | 67.1 (15) | 73.2 (14.6) | 78.5 (18.4) | 59.7 (22.7) | 70 (26.6)
  Week 4: number analyzed (Participants) | 19 | 20 | 19 | 20 | 20
  Week 4 | 49.9 (18) | 49.8 (21.1) | 55.5 (27) | 40.2 (24.1) | 52.5 (27.3)
  Week 8: number analyzed (Participants) | 19 | 20 | 18 | 20 | 20
  Week 8 | 35.9 (23.4) | 39.7 (19.5) | 47.2 (20.8) | 33 (27.2) | 39.1 (28.8)
  Week 12: number analyzed (Participants) | 17 | 20 | 19 | 19 | 18
  Week 12 | 28.7 (20.2) | 31.2 (21.6) | 36.7 (25.3) | 29.8 (29.7) | 40.4 (29)
  Week 24: number analyzed (Participants) | 17 | 18 | 17 | 20 | 20
  Week 24 | 16.9 (21) | 23.1 (25.6) | 28.5 (26) | 23.8 (28.2) | 32.1 (31.4)

2. Primary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH), Treated Subjects
Description: The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Time Frame: Baseline, 4, 8, 12, and 24 weeks
Population: Analysis conducted on patients at Baseline, 4, 8, 12, and 24 weeks time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
score on a scale
  Baseline | 43.7 (13.9) | 43.5 (13.5) | 40.1 (19.8) | 40 (15.3) | 41.3 (18.5)
  Week 4: number analyzed (Participants) | 19 | 20 | 18 | 20 | 20
  Week 4 | 29.2 (12.5) | 30.9 (12.8) | 34.1 (18.3) | 27.8 (20.2) | 38.3 (22.9)
  Week 8: number analyzed (Participants) | 19 | 20 | 18 | 20 | 20
  Week 8 | 21.8 (11.5) | 23 (14.2) | 24.7 (14.9) | 19.7 (16.4) | 25.1 (22.5)
  Week 12: number analyzed (Participants) | 17 | 20 | 19 | 19 | 18
  Week 12 | 12.6 (8.6) | 16.7 (13.2) | 19.8 (15.3) | 16.1 (15.9) | 24.5 (23.7)
  Week 24: number analyzed (Participants) | 17 | 18 | 17 | 20 | 20
  Week 24 | 7.2 (9.6) | 11.4 (9.9) | 14.5 (17.3) | 13.8 (15.6) | 19.6 (24.3)

3. Primary Outcome: Total Score Patient Rated Tennis Elbow Evaluation (PRTEE), All Treated Subjects
Description: The Pain and disability measured by the Patient Rated Tennis Elbow Evaluation (PRTEE) is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis (also known as "tennis elbow"). The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales:
  1. PAIN subscale (0 = no pain, 10 = worst imaginable)
     -Pain - 5 items
  2. FUNCTION subscale (0 = no difficulty, 10 = unable to do)
     * Specific activities - 6 items
     * Usual activities - 4 items
  In addition to the individual subscale scores, a total score can be computed on a scale of 100 (0 = no disability), where pain and functional problems are weighted equally
Time Frame: Baseline, 4, 8, 12, and 24 weeks
Population: Analysis conducted on patients at Baseline, 4, 8, 12, and 24 weeks time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
score on a scale
  Baseline: number analyzed (Participants) | 20 | 20 | 19 | 19 | 20
  Baseline | 52.6 (17.9) | 56 (14.3) | 48.3 (16.3) | 52.6 (20.7) | 52.3 (22.9)
  Week 4: number analyzed (Participants) | 19 | 20 | 19 | 20 | 20
  Week 4 | 34.7 (14.5) | 39.2 (15.3) | 39.3 (21.7) | 32.2 (23.9) | 43.4 (24.3)
  Week 8: number analyzed (Participants) | 19 | 20 | 18 | 20 | 20
  Week 8 | 25.2 (15.2) | 26.9 (17.4) | 28.9 (15.1) | 25.4 (21) | 28.6 (24.9)
  Week 12: number analyzed (Participants) | 17 | 20 | 19 | 19 | 18
  Week 12 | 13.5 (8) | 18.2 (16.4) | 22.3 (16.4) | 20.1 (22.7) | 26.8 (24.8)
  Week 24: number analyzed (Participants) | 17 | 18 | 17 | 20 | 20
  Week 24 | 7.8 (10) | 12.1 (12.4) | 16.2 (17.9) | 16.8 (19.3) | 22.3 (27.3)

4. Primary Outcome: Grip Strength Test, All Treated Subjects
Description: Grip strength testing will be performed to evaluate changes in the strength and sincerity of effort as a result of treatment for lateral epicondylitis. Testing will be performed to assess the pain-free grip strength (performing the test until discomfort is felt) and maximum grip strength (performing the test to the maximum of their ability). The test will be performed while the patient is standing with the elbow in full extension, as this position has been used to assess grip strength in patients with lateral epicondylitis. A Jamar Plus+ Digital Hand Dynamometer with the grip in the second position will be used because the second position has been assumed to be the most reliable and consistent position. Patients will be asked to perform three repetitions of each test (pain-free and maximum) at each study interval and the mean score will be calculated and used for analysis.
Time Frame: Baseline, 4, 8, 12, and 24 weeks
Population: Analysis conducted on patients at Baseline, 4, 8, 12, and 24 weeks time points.
Measure: Mean (Standard Deviation); unit: lbs.
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
lbs.
  Baseline | 42.6 (30.1) | 33.4 (24.1) | 47.6 (29.4) | 39.6 (28.9) | 39.7 (23.2)
  Week 4: number analyzed (Participants) | 19 | 20 | 19 | 20 | 19
  Week 4 | 40.2 (25.6) | 44.5 (32) | 48.3 (33) | 52 (30.2) | 41.9 (26.3)
  Week 8: number analyzed (Participants) | 19 | 20 | 17 | 20 | 20
  Week 8 | 53.5 (27.8) | 50.6 (36.3) | 64.6 (35) | 53.3 (29) | 54.8 (26.4)
  Week 12: number analyzed (Participants) | 17 | 20 | 19 | 19 | 18
  Week 12 | 58.2 (28.1) | 61 (37.7) | 67.5 (38.3) | 61.1 (32.1) | 45.1 (25.3)
  Week 24: number analyzed (Participants) | 17 | 18 | 17 | 20 | 19
  Week 24 | 66.4 (26.4) | 69.1 (37.5) | 79.9 (33.4) | 69.9 (29.1) | 62.9 (25.7)

5. Primary Outcome: Maximum Grip Strength, Treated Subjects
Description: A higher grip strength score indicates an improvement. A positive change from baseline indicates an improvement. Grip strength testing will be performed to evaluate changes in the strength and sincerity of effort as a result of treatment for lateral epicondylitis. Testing will be performed to assess the pain-free grip strength (performing the test until discomfort is felt) and maximum grip strength (performing the test to the maximum of their ability). The test will be performed while the patient is standing with the elbow in full extension, as this position has been used to assess grip strength in patients with lateral epicondylitis. A Jamar Plus+ Digital Hand Dynamometer with the grip in the second position will be used because the second position has been assumed to be the most reliable and consistent position. Patients will be asked to perform three repetitions of each test (pain-free and maximum) at each study interval and the mean score will be calculated and used for analysis.
Time Frame: Baseline, 4, 8, 12, and 24 weeks
Population: Analysis conducted on patients at Baseline, 4, 8, 12, and 24 weeks time points.
Measure: Mean (Standard Deviation); unit: lbs.
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
lbs.
  Baseline | 60.4 (35) | 58.7 (33.1) | 71.8 (38.9) | 60.3 (31.2) | 61.3 (29.7)
  Week 4 | 62.9 (26.2) | 63.5 (33.1) | 64.2 (37.2) | 68.9 (35.5) | 62 (33)
  Week 8 | 73.3 (29.3) | 66.4 (31.3) | 72.9 (37) | 71.6 (30) | 66.9 (31.5)
  Week 12 | 78.9 (29.9) | 68.6 (31.2) | 81.8 (39.7) | 74.5 (32.8) | 65.1 (30)
  Week 24 | 82.5 (32.7) | 71 (32.5) | 80.7 (33.7) | 77.8 (27) | 76.4 (30.9)

ADVERSE EVENTS:
Time Frame: Patients were assessed through study completion scheduled at 24 weeks following surgery.
Arm/Group | Placebo Control | 0.45 mg rhPDGF-BB | 0.75 mg rhPDGF-BB | 1.5 mg rhPDGF-BB | 3.0 mg rhPDGF-BB
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 2/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 15/20 | 20/20 | 18/20 | 16/20 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Control (N=20) | 0.45 mg rhPDGF-BB (N=20) | 0.75 mg rhPDGF-BB (N=20) | 1.5 mg rhPDGF-BB (N=20) | 3.0 mg rhPDGF-BB (N=20)
Injection site calcification (General disorders) | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Control (N=20) | 0.45 mg rhPDGF-BB (N=20) | 0.75 mg rhPDGF-BB (N=20) | 1.5 mg rhPDGF-BB (N=20) | 3.0 mg rhPDGF-BB (N=20)
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site calcification (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site coldness (General disorders) | 1 | 0 | 0 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 1 | 0 | 2
Injection site haematoma (General disorders) | 0 | 1 | 1 | 1 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 1
Injection site inflammation (General disorders) | 0 | 1 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 0 | 2 | 1
Injection site pain (General disorders) | 3 | 8 | 5 | 6 | 12
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 6 | 1 | 3 | 4
Injection site warmth (General disorders) | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 2
Tenderness (General disorders) | 0 | 0 | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Conjunctival abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 7 | 4 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Renal function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 9 | 4 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 2 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 2 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 2 | 6
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 2 | 0 | 0 | 4
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Adjustment disorder with anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 4
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Female sterilisation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0
Uterine dilation and curettage (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
While this preliminary study suggests similar safety profiles for PDGF and placebo, future studies with larger sample sizes, possibly different concentrations, and tighter inclusion criteria are needed to definitely assess the effectiveness of PDGF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes